CLINICAL TRIAL: NCT05902650
Title: Correlation of Biochemical Indexes and Retinal Hemodynamic in Patients With Different Degrees of Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mingzhe Cao (Other)
Responsible Party: Sponsor-Investigator, Mingzhe Cao, Attending ophthalmologist, The Seventh Affiliated Hospital of Sun Yat-sen University
Organization: The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Other Study IDs: MCao
Record Dates: First submitted 2023-06-01; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: diabetic patients with no diabetic retinopathy
  Interventions: Diagnostic Test: imaging
- Group 2: diabetic patients with mild nonproliferative diabetic retinopathy
  Interventions: Diagnostic Test: imaging
- Group 3: diabetic patients with moderate and severe nonproliferative diabetic retinopathy
  Interventions: Diagnostic Test: imaging
- Group 4: diabetic patients with proliferative diabetic retinopathy
  Interventions: Diagnostic Test: imaging

INTERVENTIONS:
Diagnostic Test: imaging — imaging

SUMMARY:
All OCTA data and biochemical indexes of diabetic patients were acquired. A prediction model of diabetic retinopathy was built, and the random forest method was used to identify sensitive indicators.

DETAILED DESCRIPTION:
Diabetic patients at the Department of Ophthalmology of the Seventh Affiliated Hospital of Sun Yat-sen University were selected as research participants. All OCTA data and biochemical indexes were acquired. A prediction model of diabetic retinopathy was built, and the random forest method was used to identify sensitive indicators.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes

Exclusion Criteria:

* various other types of retinal and choroidal disease;
* history of any intraocular surgery or treatment (including intravitreal injection, retinal photocoagulation etc.
* with severe refractive medium opacity that could affect fundus examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
fasting blood glucose (FBG) | the time of the patient's first 1 day visit
  biochemical indexes
glycosylated hemoglobin (HbAlc) | the time of the patient's first 1 day visit
  biochemical indexes
OCTA data | the time of the patient's first 1 day visit
  An image of the 3mm×3mm and 6 mm×6 mm macular areas detected by OCTA were captured. Quantitative analysis of vascular density and perfusion density of superficial capillary plexus in the macular area were automatically calculated using built-in software on the device.

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhe Cao, Principal Investigator — The Seventh Affiliated Hospital of Sun Yat-sen University
Locations (1):
- The Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The research has not been completed.